CLINICAL TRIAL: NCT05483426
Title: Prevalence of Sexual Addiction in an Inmate Population at the Muret Detention Center in Haute-Garonne.
Brief Title: Prevalence of Sexual Addiction in an Inmate Population at the Muret Detention Center in Haute-Garonne (PAS-CD)
Acronym: PAS-CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federation Regionale de Recherche en Psychiatrie et Sante Mentale Occitanie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00342-41
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Sexual Addiction
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interviews (Other): semi-directive interview
  Interventions: Other: semi-structured Interviews

INTERVENTIONS:
Other: semi-structured Interviews — semi-structured interview conducted by a psychiatrist

SUMMARY:
Sexual addiction, also known as hypersexuality or compulsive sexuality, is a human sexual behavior that results in a continuous and persistent search for sexual pleasure. Replacing the former terms satyriasis and nymphomania, the World Health Organization (WHO) ICD-11 has referred to this disorder as "compulsive sexual behavior disorders".

From multiple causes (iatrogeny, neurological causes, psychiatric causes, psychopathological hypotheses), but still only partially known, the inclusion of this disorder among impulsivity-related disorders, obsessive-compulsive disorders or addiction-related disorders is still debated in the scientific literature. Thus, in the absence of sufficient robust scientific data, DSM-5 refused to include this disorder in its classification.

However, the consequences of this disorder on the psychosocial functioning of individuals are not negligible, which can go as far as the precipitation of a transition to an heteroaggressive act which can thus lead to incarceration.

The prevalence of this disorder in the general population is estimated between 2 and 6% based on current literature data. This rate appears to be higher among men and more specifically among sex offenders.

However, some authors have noted that the difficulty in determining a clear prevalence of sexual addiction may be related to the still poorly defined diagnostic criteria for this disorder as well as the choice of measurement tools.

In the inmate population, to our knowledge, there are no French prevalence studies of this disorder. In addition, no studies have been conducted to compare the prevalence of sexual addiction among sex offenders (SASO) with that among non-sex offenders (SANSO).

We hope that better screening for addiction would enable better management of patients with this disorder, promoting their psychosocial rehabilitation and well-being, so as to prevent the recurrence of a transition to sexual arousal.

DETAILED DESCRIPTION:
This study is intended to assess the prevalence of sexual addiction among a population of detainees at the Muret detention center in Haute-Garonne.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Detainees at Muret Detention Center
* Aged between 18 and 65 at the time of the search
* And having agreed to participate in the research.

Exclusion Criteria:

* Person under legal protection, guardianship or curatorship ;
* Insufficient command of the French language
* Existence of cognitive disorders preventing a good understanding of the information relating to the study or the various questionnaires.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The main objective is to determine the prevalence of sexual addiction among a population of men incarcerated at the Muret detention center in Haute-Garonne. | Day 1
  The primary endpoint is the presence of a patient's sexual addiction defined by a score greater than 13 on the Carnes screening test.

SECONDARY OUTCOMES:
Determine the prevalence of sexual addiction in a population of sexual offenders | Day 1
  The distribution of the proportions of people with sexual addiction is defined by a score greater than 13 on the Carnes screening test in two population groups, perpetrators of sexual offenses and perpetrators of non-sexual offenses.
Determine the prevalence of sexual addiction in a population of non-sexual offenders | Day 1
  The distribution of the proportions of people with sexual addiction is defined by a score greater than 13 on the Carnes screening test in two population groups, perpetrators of sexual offenses and perpetrators of non-sexual offenses.
Compare the prevalence of sexual addiction in these two populations | Day 1
  The distribution of the proportions of people with sexual addiction is defined by a score greater than 13 on the Carnes screening test in two population groups, perpetrators of sexual offenses and perpetrators of non-sexual offenses.
Determine any addictive and psychiatric co-morbidities associated with each population | Day 1
  The presence of psychiatric disorders is defined using the Mini International Neuropsychiatric Interview (MINI) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Julien DA COSTA, Toulouse, France

IPD SHARING:
Plan to Share IPD: No